CLINICAL TRIAL: NCT00874562
Title: Rapamycin in Relapsed Acute Lymphoblastic Leukemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Brigham and Women's Hospital (Other); Boston Children's Hospital (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Lewis B. Silverman, M.D., Principal Investigator, Dana-Farber Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 06-429
Record Dates: First submitted 2009-04-01; First posted 2009-04-02 (Estimated); Last update posted 2016-11-23 (Estimated); Status verified 2016-11

CONDITIONS: Acute Lymphoblastic Leukemia
Keywords: rapamycin; corticosteroid; ALL
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Adrenal Cortex Hormones; Sirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Steroid Only (Active Comparator): Corticosteroid Alone
  Interventions: Drug: Corticosteroid
- Steroid plus Rapamycin (Active Comparator): Corticosteroid plus Rapamycin
  Interventions: Drug: Corticosteroid; Drug: Rapamycin

INTERVENTIONS:
Drug: Corticosteroid — Initial dose of corticosteroid given intravenously. After the first dose, corticosteroid will be taken orally every 8 hours for the duration of the five-day period
Drug: Rapamycin — Taken orally mixed with water or orange juice
  Other Names: sirolimus
  Arms: Steroid plus Rapamycin

SUMMARY:
This is a research study designed to look at the biological effects of two drugs on leukemia cells. In this study, we are comparing the effects of drugs called corticosteroids when used alone or with another drug called rapamycin. Rapamycin is a drug that prevents the body's immune system from working normally. It has been used for many years after kidney transplants to prevent rejection of the organ. Recent work suggests that rapamycin may also help treat leukemia and other cancers.

DETAILED DESCRIPTION:
* Participants will be randomized into two groups; one group will receive corticosteroid alone, and the other group will receive rapamycin and corticosteroid.
* The length of treatment will be 5 days, during which time we will collect blood samples to measure the biologic effects of these drugs. Because these drugs will be given for a short period of time only, this study is not designed to treat or cure the participants leukemia. After the 5-day period, participants may resume other cancer-directed therapies.

ELIGIBILITY:
Inclusion Criteria:

* Documented acute lymphoblastic leukemia (L1 or L2 subtypes)
* First or subsequent relapse
* 365 days of age or older
* Greater than 7 days from any chemotherapy or immunotherapy, with the exception of intrathecal chemotherapy
* Absolute peripheral leukemia blast count of 1000 cells/ul or greater
* Patient (or parent/guardian if patient is less than 18 years of age) must sign informed consent

Exclusion Criteria:

* Burkitts leukemia (acute lymphoblastic leukemia L3 subtype)
* Uncontrolled active infection
* Pregnancy or mothers who are nursing
* Patient currently taking rapamycin
* Patients with significant liver dysfunction as outlined in protocol
* Severe concurrent disease, which in the judgment of the investigator, would make the patient inappropriate for entry into the study
* Active psychiatric disease, substance abuse, or mental illness that would interfere with cooperation with the requirements of the trial

Min Age: 365 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2007-07; Primary Completion 2009-11 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Compare changes in gene expression signatures in steroid alone versus steroid plus rapamycin treated patients. | 3 years
Compare biologic measures of "pro-apoptotic state" in steroid alone versus steroid plus rapamycin treated patients | 3 years

SECONDARY OUTCOMES:
Assess clinical response by percent reduction of peripheral leukemia blasts at day 2 of therapy and at completion of the 5-day investigational window | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Lewis Silverman, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana-Farber Cancer Institute, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No